CLINICAL TRIAL: NCT06387654
Title: Constitution of a Collection of Biological Samples With the Aim of Carrying Out Clinico-biological and Physiopathological Investigations of Autoimmune, Dysimmune or Auto-inflammatory Dermatological Diseases
Brief Title: Clinico-biological Collection of Autoimmune, Dysimmune or Auto-inflammatory Dermatological Diseases
Acronym: TekAPo
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0361
Record Dates: First submitted 2024-03-28; First posted 2024-04-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Bullous Dermatosis; Dysimmune Dermatological Diseases; Auto-inflammatory Dermatological Diseases; Skin Diseases
Keywords: auto-inflammatory dermatological diseases; Cutaneous lupus; scleroderma; dermatomyositis; psoriasis; eczema; new therapies
MeSH Terms: conditions — Skin Diseases; Scleroderma, Diffuse; Dermatomyositis; Psoriasis; Eczema | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, CSF, saliva, stool, urine, other body fluids and tissue biopsies, hair follicles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suffering from autoimmune, dysimmune or auto-inflammatory dermatological disease: Biological samples will be collected in the normal diagnosis and follow-up process
  Interventions: Biological: Blood sampling; Biological: Remainders of samples taken as part of the treatment

INTERVENTIONS:
Biological: Blood sampling — Blood will be taken in larger quantity
Biological: Remainders of samples taken as part of the treatment — blood, CSF, saliva, stools, urine, other biological fluids and tissue biopsies, hair follicles

SUMMARY:
The aim of this project is to start a biological and clinical collection of patients presenting autoimmune, dysimmune or auto-inflammatory dermatological diseases. This collection will provide appropriate biological samples to identify new biomarkers and to be accessible to the medical, scientific and industrial communities for the identification of new therapeutic strategies.

DETAILED DESCRIPTION:
Autoimmune diseases include around a hundred different clinical entities which are for the most part rare pathologies but which, in combination, concern 5-8% of the adult population with a strong female predominance (FAI²R: the disease chain rare autoimmune and auto-inflammatory drugs, fai2r.org). The common denominator of all these diseases is based on the breakdown of self-tolerance which is the origin of self-reactivity and whose physiopathological mechanisms are still not fully understood, which generates numerous cross-sectional or fundamental studies. In addition to this complexity, there are significant inter-individual variabilities which lead to the definition of subgroups of patients on the basis of the clinical-biological profile and / or the response to treatments. Consequently, and in view of the need to establish the diagnosis early and then to propose the best treatment in the perspective of an individualized medicine, the clinical, biological and genetic characteristics of these subgroups of patients must be explored in order to improve diagnostic and therapeutic capacities.

ELIGIBILITY:
Inclusion Criteria:

Skin damage of documented or probable autoimmune, dysimmune or autoinflammatory origin.

The patients included may be adults or children, and will be:

* Patients with autoimmune bullous dermatoses (pemphigus, pemphigoid and others),
* Patients with systemic autoimmune diseases associated with skin damage (lupus, scleroderma, dermatomyositis for example),
* Patients with cutaneous lupus
* Patients with dysimmune skin diseases (psoriasis, eczema)
* Patients with immuno-induced dermatological disorders or drug dermatitis
* Patients receiving, or likely to receive, new, innovative therapies (new molecule on the market, checkpoint inhibitors, gene therapy, cell therapy, etc.).

Patients with dermatological damage whose autoimmune, dysimmune or auto-inflammatory origin is suspected

Exclusion Criteria:

* Patients under protective supervision (guardianship, curators)
* Patients under 6 years old
* Pregnant or breastfeeding woman

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune, dysimmune or auto-inflammatory dermatological disease
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Building a collection of biological samples and clinical-biological data from patients with autoimmune, dysimmune or auto-inflammatory dermatological disease | Day 0 and through study completion, an average of 1 year
  Blood sampling

SECONDARY OUTCOMES:
Identification of new autoantibodies | Day 0 and through study completion, an average of 1 year
  Western blot or immunoprecipitation method
Identification of biomarkers regarding the severity (such as cytokines, survival factors) in order to help the therapeutic decisions | Day 0 and through study completion, an average of 1 year
  Proteomic analysis of sera and plasma samples at diagnosis and during follow up
Exploration of the pathophysiological mechanisms of rare autoimmune dermatological pathologies | Day 0 and through study completion, an average of 1 year
  Knock-out or knock-in animal models for one specific protein will be used to determine in vivo if the pathophysiological mechanisms of Dermatological Diseases can be induced by the abnormal expression of this protein.
  Analysis of the phenotypic profiling of blood immune cells by multicolor fluorescence-activated cell sorter (FACS) analysis and of the transcriptomic profiling of blood immune cells by RNA sequencing
Comparison of blood cells populations determinants with flow cytometry, before and after cell therapy and in patients responder or not responder to cell therapy | Day 0 and through study completion, an average of 1 year
  Exploring blood cell populations before and after cell therapy with flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Chloé BOST, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No